CLINICAL TRIAL: NCT06674356
Title: The Effects of Chin Tuck Against Resistance Exercise on Swallowing Function, Depression, and Quality of Life in Acute Stroke Patients With Dysphagia
Brief Title: The Effects of Chin Tuck Against Resistance Exercise on Acute Stroke Patients With Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202408146RINB
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Acute Stroke; Dysphagia
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group:Participants in this group will receive traditional swallowing rehabilitation combined with chin tuck against resistance (CTAR) training to enhance suprahyoid muscle strength and improve swallowing function.
  Interventions: Behavioral: chin tuck against resistance exercise
- Control Group (Placebo Comparator): Control Group:Participants in this group will receive only traditional swallowing rehabilitation without any additional CTAR training.
  Interventions: Behavioral: chin tuck against resistance exercise

INTERVENTIONS:
Behavioral: chin tuck against resistance exercise — Both groups of patients will receive traditional swallowing rehabilitation therapy; however, the experimental group will additionally perform CTAR exercises. The procedure is as follows:Ask the patient to sit, then, press the chin firmly against the inflatable rubber ball, for isometric exercise, the chin is pressed down against the resistance of the ball and held for 60 seconds as one round, with a total of three rounds. And for isotonic exercise, the chin presses down against the resistance of the ball and holds for one second per repetition, with a total of 30 repetitions. Performing both isometric and isotonic exercises constitutes one set of exercises.
  For isometric exercise, the chin is pressed down against the resistance of the ball and held for 60 seconds as one round, with a total of three rounds. For isotonic exercise, the chin presses down against the resistance of the ball and holds for one second per repetition, with a total of 30 repetitions.
  Other Names: Traditional swallowing rehabilitation

SUMMARY:
The aim of this study is to investigate the effects of chin tuck against resistance exercise on swallowing function, depression, and quality of life in acute stroke patients with dysphagia.

DETAILED DESCRIPTION:
The study is an experimental research design, with participants randomly assigned to either the experimental group or the control group. The experimental group will undergo chin tuck against resistance exercises, while the control group will receive traditional swallowing rehabilitation training. The subjects of this study are patients from the neurology and rehabilitation wards of a medical center in northern Taiwan. The research tools include a personal basic information questionnaire, the standardized swallowing assessment, the Functional Oral Intake Scale, the Patient Health Questionnaire-9, and the Taiwan version of the Swallowing Quality of Life Questionnaire. Data collection for both groups will be conducted using a pre-test and post-test method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with hemorrhagic or ischemic stroke, including those with initial diagnoses or recurrent strokes.
2. Patients who did not pass the swallowing screening based on the standard swallowing scale.
3. Adults aged 18 years and older.
4. Vital signs are stable: systolic blood pressure (hemorrhagic < 160 mmHg, ischemic < 220 mmHg), heart rate 40-130 beats per minute, and oxygen saturation > 92%.
5. The patient's consciousness is clear, able to express themselves, can communicate in Mandarin or Taiwanese, and can follow commands to perform actions.
6. The patient can be in a seated position.

Exclusion Criteria:

1. Patients who have had a stroke for more than one month (inclusive).
2. Patients with a history of depression or related mental health disorders.
3. Patients with a history of neck pain, injury, or disease.
4. Patients who have previously undergone tracheostomy or have a tracheostomy tube in place.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-12-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
swallowing function | before intervention and up to 6 weeks
  Use the Functional Oral Intake Scale(FOIS) 、calculating the residual volume of 60 ml of water, swallowing speed, and whether a nasogastric tube is in place to assess swallowing function. FOIS items range from 1 to 7，the higer the better swallowing function。The less residual water and fast swallowing speed(ml/sec), the better the swallowing function. The absence of a nasogastric tube also indicates improvement in swallowing.

SECONDARY OUTCOMES:
Depression | before intervention and up to 6 and 10 weeks
  Use the Patient Health Questionnaire(PHQ-9) to assess depression，the score ranges from 0 to 27 points: 0-4 indicates no depressive symptoms, 5-9 indicates mild depression, 10-14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Swallowing-Related Quality of Life | before intervention and up to 6 and 10 weeks
  use the Taiwanese version of the Swallowing Quality of Life Questionnaire to evaluate quality of Life. The questionnaire consists of 44 questions, scored on a 5-point Likert scale. Each question has a maximum score of 5 and a minimum score of 1. Higher scores on the questionnaire indicate a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nursing, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No